CLINICAL TRIAL: NCT01185977
Title: Biomarkers of Antidepressant Treatment in Adolescents With Major Depression
Brief Title: Biomarkers of Antidepressant Treatment in Adolescents With Major Depression (The Adolescents MDD Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ian A. Cook, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 090713201
Record Dates: First submitted 2010-04-06; First posted 2010-08-20 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Fluoxetine; QEEG; cordance; ATR
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoxetine (Active Comparator): 1 week single-blinded placebo lead-in and double-blinded FLX treatment for 8 weeks
  Interventions: Drug: Fluoxetine
- Placebo (PBO) (Placebo Comparator): Placebo treatment for 9 weeks of study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — one-week single-blind PBO-lead-in phase, FLX 10 mg/d for 4 days then 20 mg/d of FLX thereafter
  Arms: Fluoxetine
Drug: Placebo — One pill of PBO for 4 days then two pills of PBO thereafter
  Arms: Placebo (PBO)

SUMMARY:
This study will aim to evaluate the use of Electroencephalography (EEG) biomarkers in adolescent depression. Two specific hypotheses will be tested:

H1: Early decreases in prefrontal cordance values will be greater in responders to antidepressant therapy than in medication non-responders.

H2: Subjects with high Antidepressant Treatment Response(ATR) Index values [i.e., predicted to show symptomatic improvement with fluoxetine (FLX)] will achieve greater improvement in symptoms and in functional status than those with low ATR values.

Exploratory analyses will be undertaken to compare and contrast the cordance changes and ATR values in medication and placebo-treated responders and non-responders.

DETAILED DESCRIPTION:
A total of 26 adolescent subjects with Major Depressive Disorder(MDD), ages 12 to 20, will be consented and join this project at UCLA. For analytic purposes, we will define an "enrolled" subject as one who has completed the single-blind lead-in week and one week of double-blind treatment, and the three EEG recordings at these visits, as any subject who leaves the project prior to that point cannot contribute useful data to testing our hypotheses.

Subjects who enroll in this project will receive 1 week of single-blind placebo lead-in, followed by 8 weeks of double-blind randomized treatment either with fluoxetine (FLX), a Selective Serotonin Reuptake Inhibitor (SSRI) with FDA approval for use in this age group, or with placebo. Brain activity will be assessed with Qualitative EEG (QEEG) recording at pretreatment baseline, after lead-in, and at 1, 2, 4, and 8 weeks of treatment to expand the evidence base on the neurophysiology of treatment response in adolescents. Subjects will be assessed for symptom change, adverse events, and suicidality at each visit. Functional measures related to treatment will be assessed at baseline and at weeks 4 and 8. Subjects and the staff who interact with them will be blinded to QEEG biomarker values during the project.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with non-psychotic, unipolar Major Depressive Disorder (MDD) based on the K-SADS-PL
* A score of ≥ 45 on the Children's Depression Rating Scale-Revised (same threshold as TADS). As with the TADS trial, depressed mood must have been present in at least 2 of 3 contexts (home, school, among peers) for at least 6 weeks prior to consent.
* Age range: 14-18.
* Patients with suicidal ideation are eligible only if the thoughts of death or of life not being worth living are not accompanied by a plan or intention for self-harm.

Exclusion Criteria:

* Subjects will have no unstable medical illness that would prevent completion of participation in the trial (determined as needed from physical examination, ECG, laboratory safety tests, as well as a review of systems). Other specific exclusionary criteria also are based on the BRITE-MD parameters, and include:

  1. mentally or legally incapacitated, unable to give informed consent;
  2. meets DSM-IV criteria for anorexia nervosa, bulimia nervosa, obsessive-compulsive disorder, any cognitive disorder, bipolar disorder, psychotic disorder, or major depression with psychotic features;
  3. MMSE (Folstein et al., 1975) score ≤ 24;
  4. evidence of drug dependency or substance abuse within the preceding nine months;
  5. stable and in remission on current psychotropic medication(s);
  6. any ECT within the past six months;
  7. failure to tolerate FLX or treatment failure with an adequate trial of FLX in the current episode;
  8. FLX would be contraindicated (e.g., hyponatremia with a prior SSRI);
  9. treatment with an MAOI within the past four weeks;
  10. any medical illness severe enough to significantly affect brain function or to interfere with interpretation of study results;
  11. history of seizures, brain surgery, skull fracture, significant head trauma, or abnormal EEG;
  12. psychiatric hospitalization indicated (e.g., imminent danger to self or others);
  13. initial QEEG recording is contaminated with artifact so that determination of the biomarker is precluded;
  14. use of medications known to affect brain function (e.g., antidepressants, anticonvulsants/mood stabilizers, anticholinergics, antipsychotics, benzodiazepines - same list as in BRITE-MD). Based on the TADS trial, we will also exclude for concurrent diagnoses of attention-deficit hyperactivity disorder managed with psychostimulants, pervasive developmental disorder, and mental retardation (mild, moderate, severe, or profound);
  15. subject is currently pregnant, or is of child-bearing potential and not using a medically acceptable means of birth control (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Score on Children's Depression Rating Scale-Revised | Measured over 8 weeks

SECONDARY OUTCOMES:
Score on Hamilton Depression Rating Scale (HAM-D) | Measured over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Cook, MD, Principal Investigator — Universityof California Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- See also: Related Info — http://www.DepressionLA.com